CLINICAL TRIAL: NCT03013192
Title: Effect of a Three Month Automated Messaging Intervention on Patient Compliance to Physical Therapy Regimens and on Clinical Outcomes
Brief Title: Three Month Automated Messaging Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB and institutional re-assessment
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Scott Kaar, MD, Associate Professor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27655
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Rotator Cuff Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No text message reminders, usual patient protocol
- Intervention (text messaging) (Experimental): Text message reminders for PT
  Interventions: Other: Text message reminder

INTERVENTIONS:
Other: Text message reminder — Patients will receive automated text message reminders regarding their physical therapy
  Arms: Intervention (text messaging)

SUMMARY:
Patients who are prescribed physical therapy exercises for their shoulder will have increased compliance to their PT exercises, an increased ASES score, and will have increased range of motion (or reach maximum range of motion earlier) at the end of the 3 month EpxPhysicalTherapy intervention.

DETAILED DESCRIPTION:
Patient compliance to their prescribed physical therapy (PT) exercises is reported to be 22-40% in various studies. Further, Vasey et al. found that about 8% of patients do not even schedule a follow up PT appointment after it is prescribed. Low adherence presents a problem since long term completion of prescribed home exercises has been correlated with improved health outcomes. Sluijs et al. found that low adherence to PT exercises can be primarily attributed to three factors: (1) the barriers patients perceive and encounter, (2) the lack of positive feedback, and (3) the degree of helplessness. An automated phone/texting system can help with these three points by increasing positive feedback, increasing compliance, and monitoring patient progress. The system can continually remind the patient that their end goal is possible, which will decrease their feeling of helplessness in their condition.

Provide an introduction and background information. Describe past experimental and/or clinical findings leading to the formulation of the study, if applicable. Investigator Initiated studies must cite references in the response provided or attach a bibliography. *?HELP?*

Patient compliance to their prescribed physical therapy (PT) exercises is reported to be 22-40% in various studies [1-4]. Further, Vasey et al. found that about 8% of patients do not even schedule a follow up PT appointment after it is prescribed [5]. Low adherence presents a problem since long term completion of prescribed home exercises has been correlated with improved health outcomes. Sluijs et al. found that low adherence to PT exercises can be primarily attributed to three factors: (1) the barriers patients perceive and encounter, (2) the lack of positive feedback, and (3) the degree of helplessness [2]. An automated phone/texting system can help with these three points by increasing positive feedback, increasing compliance, and monitoring patient progress. The system can continually remind the patient that their end goal is possible, which will decrease their feeling of helplessness in their condition.

The American Shoulder and Elbow Surgeons (ASES) created a survey form that evaluates the shoulder function of a patient. The survey is scored out of 100 points (100 being best possible shoulder function and 0 being worst possible shoulder function). The form can be filled out on an iPad online, and the score recorded by a member of the medical team. This screening form has been validated by numerous studies, and has been specifically validated for patients with non-operative rotator cuff pain/abnormalities (the population that this study is proposing to study).

Telemedicine shows promise in improving the outcomes of orthopedic interventions. Medication adherence and patient outcomes have been shown to improve in interventions that include reminders. Also, because the adoption of cell phones is nearly ubiquitous worldwide and the vast majority of cell phone users text message, a text-message-based intervention seems particularly promising.

Many studies have shown that SMS text messaging has increased treatment compliance. PT adherence to prescribed exercises seems to be limited by compliance, so Epharmix along with several orthopedic surgeons set out to develop an intervention. The result, EpxPhysicalTherapy (EpxPT), is an automated system that ensures that patients have both scheduled their physical therapy appointment and have performed their home exercises. It also sends motivational text messages to the patient to encourage the participant to perform their exercises since a lack of positive reinforcement has been correlated with decreased compliance. When a patient identifies that they have been unable to schedule a PT appointment or have not completed their exercises for multiple days in a row, an alert is sent to the healthcare team.

The system was designed to deliver either voice or text-based automated messages to patients in a way that avoids an additional burden on the healthcare team. EpxPT offers numerous advantages to strictly app-based or text message-based systems in both older and underprivileged patient populations. Older patients, who may be more comfortable with voice messages, have that option, and patients without a smartphone will still be able to receive the intervention.

Patients identified to be eligible for this study and have consented will be randomly assigned to one of two groups: Group 1 will receive the standard of care alone (control) and Group 2 will receive the EpxPT intervention. In Group 2, EpxPT will remind the patient to schedule their first PT appointment. Group 2 patients will also be asked if they have completed their prescribed PT exercises every other day. They will then be sent a motivational text messages or voice call in order to highlight the importance of completing their PT regimen. Group 2 patient compliance will be tracked through the text responses recorded in the Epharmix database. Both Group 1 and Group 2 patients will be seen at a follow up appointment once a month for three months. At this appointment, patients in both groups will be asked about their PT compliance (this will be the measurement of compliance for Group 1), and range of motion and a ASES score will be measured.

* Aim 1: To compare control and intervention group compliance to their prescribed physical therapy home exercise regimen
* Aim 2: To compare control and intervention group shoulder range of motion after a 3 month intervention
* Aim 3: To compare control and intervention group ASES scores after a 3 month intervention

ELIGIBILITY:
Inclusion Criteria:

* Anterior or lateral shoulder tenderness
* Positive clinical signs of rotator cuff impingement
* X-ray with no fractures, glenohumeral arthritis, or dislocation
* Prescribed shoulder PT for their shoulder

Exclusion Criteria:

* None

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Compliance with PT | 3 months

SECONDARY OUTCOMES:
American Shoulder And Elbow Surgeons Score | 3 months
Shoulder range of motion | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No